CLINICAL TRIAL: NCT05531006
Title: Anesthesia Preferences in the COVID-19 Pandemic: General Anesthesia or Regional Anesthesia?
Status: Completed | Type: Observational
Sponsor: Erol Olcok Corum Training and Research Hospital (Other)
Responsible Party: Principal Investigator, HULYA TOPCU, Asist. Prof. M.D., Erol Olcok Corum Training and Research Hospital
Other Study IDs: Hitit Universty
Record Dates: First submitted 2022-09-03; First posted 2022-09-07 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: COVID-19; Regional anesthesia; General anesthesia
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- pandemic time group: The surgeries performed during the COVID-19 pandemic and the anesthesia techniques applied for these surgeries
  Interventions: Other: retrospective cohort study
- normal time group: The surgeries performed during the non-pandemic period and the anesthesia techniques applied in these surgeries
  Interventions: Other: retrospective cohort study

INTERVENTIONS:
Other: retrospective cohort study — retrospective patient file review

SUMMARY:
As the COVID-19 pandemic continues, humanity has started to adapt to it. In our study, we aimed to examine the adaptation of anesthetists to the pandemic and its behavioral reflection on their work.

DETAILED DESCRIPTION:
All surgeries and anesthesia methods performed in the university hospital were examined. The cases and anesthesia practices of the departments were examined. Years with and without pandemics were compared.

ELIGIBILITY:
Inclusion Criteria:

* all operations

Exclusion Criteria:

* those who refuse to have surgery
* non-operational

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The number of operations in the hospital and the anesthesia methods applied to the operations were examined retrospectively.
  Anesthesia application preferences were compared between the COVID-19 pandemic period and the non-pandemic period.
Sampling Method: Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2021-06-03 (Actual); Primary Completion 2022-12-10 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Anesthesia Preferences in the COVID-19 Pandemic: General or Regional Anesthesia? | 1 year
  number of operations and number of anesthesia methods

CONTACTS AND LOCATIONS:
Locations (1):
- Hulya TOPCU, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No